CLINICAL TRIAL: NCT05201625
Title: Markers of Severity in Covid 19 Patients
Brief Title: Markers of Severity (CD177,S100A8 &S100A12) in Sever Acute Respiratory Syndrome Coronavirus 2(SARS-COV-2) Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mai Hamdy Hamed, Assistant lecturer of microbiology and immunology in sohag general hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-21-11-22
Record Dates: First submitted 2022-01-03; First posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Active Comparator): Healthy control group
  Interventions: Diagnostic Test: real time PCR
- ICU COVID 19 patients (Active Comparator): ICU COVID 19 patients
  Interventions: Diagnostic Test: real time PCR
- non-ICU covid 19 patients (Active Comparator): non-ICU covid 19 patients
  Interventions: Diagnostic Test: real time PCR

INTERVENTIONS:
Diagnostic Test: real time PCR — real time PCR

SUMMARY:
Patients infected with covid-19 have a series of clinical manifestations, including fever, cough, myalgia or fatigue, dyspnea, even acute respiratory distress syndrome (ARDS), acute cardiac injury and secondary infection, and a lot of sever patients had to been admitted to the intensive care unit (ICU)

One of the hallmark of COVID 19 is the cytokine storm that provokes primarily pneumonia followed by systemic inflammation. besides the positive viral nucleic acid analysis and the representative pulmonary CT findings (bilateral distribution of patchy shadows and ground glass opacity), most individual patients showed the changes in several immunological and biological markers . CD177 which is one of the most clinically important neutrophil alloantigen because: i) it is a neutrophil-specific marker representative of neutrophil activation, ii) it was the most highly differentiated expressed gene in patients, and iii) the protein can be measured in the serum, making its use as a marker clinically applicable. It is expressed on neutrophils, neutrophilic metamyelocytes, and myelocytes . Given the contribution of the neutrophil activation pathway in the clustering of COVID-19 patients, neutrophil-activation features that could act as possible reliable markers of disease evolution.

ELIGIBILITY:
Inclusion Criteria:

* COVID 19 hospitalized patients (diagnosed by RT-PCR)

Exclusion Criteria:

* Age below 18 years and above 80.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Markers of severity(CD177) in Sever respiratory syndrome coronavirus 2 (SARS-COV-2) patients | one year
  - Measuring gene expression for CD 177 by RT-PCR and also by ELISA.
  Measuring gene expression for CD 177 by RT-PCR and also by ELISA.
Markers of severity(S100A8&S100A12) in Sever respiratory syndrome coronavirus 2 (SARS-COV-2) patients | one year
  Measuring level of S100A8 and S100A12 by ELISA.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Lucas C, Wong P, Klein J, Castro TBR, Silva J, Sundaram M, Ellingson MK, Mao T, Oh JE, Israelow B, Takahashi T, Tokuyama M, Lu P, Venkataraman A, Park A, Mohanty S, Wang H, Wyllie AL, Vogels CBF, Earnest R, Lapidus S, Ott IM, Moore AJ, Muenker MC, Fournier JB, Campbell M, Odio CD, Casanovas-Massana A; Yale IMPACT Team; Herbst R, Shaw AC, Medzhitov R, Schulz WL, Grubaugh ND, Dela Cruz C, Farhadian S, Ko AI, Omer SB, Iwasaki A. Longitudinal analyses reveal immunological misfiring in severe COVID-19. Nature. 2020 Aug;584(7821):463-469. doi: 10.1038/s41586-020-2588-y. Epub 2020 Jul 27. PMID 32717743
- [Background] Ong EZ, Chan YFZ, Leong WY, Lee NMY, Kalimuddin S, Haja Mohideen SM, Chan KS, Tan AT, Bertoletti A, Ooi EE, Low JGH. A Dynamic Immune Response Shapes COVID-19 Progression. Cell Host Microbe. 2020 Jun 10;27(6):879-882.e2. doi: 10.1016/j.chom.2020.03.021. Epub 2020 Apr 30. PMID 32359396